CLINICAL TRIAL: NCT04866238
Title: The Effectiveness of Clear Aligners vs Fixed Appliances on Oral Health-related Quality of Life in Patients With Severe Crowding: A 12-months Randomized Controlled Clinical Trial
Brief Title: Comparison of Oral Health Related Quality of Life Changes Between Clear Aligners and Vestibular Fixed Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-04-2021
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Teeth Crowding
Keywords: Clear aligners; Oral health related quality of life; Orthodontic; Vestibular fixed appliances; Oral health impact profile
MeSH Terms: conditions — Crowding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular fixed appliances (Active Comparator): Adult patients in this group will be treated using fixed appliances.
  Interventions: Device: Vestibular fixed appliances
- Clear aligners (Experimental): Adult patients in this group will be treated using clear aligners.
  Interventions: Device: Clear aligners

INTERVENTIONS:
Device: Vestibular fixed appliances — The fixed appliances will be applied in class1 malocclusion patients who have dental crowding, then they will be followed up for 12 months.
  Arms: Vestibular fixed appliances
Device: Clear aligners — The clear aligners will be applied in class1 malocclusion patients who have dental crowding, then they will be followed up for 12 months.
  Arms: Clear aligners

SUMMARY:
Patients who have severe crowding that required four premolars extraction will be treated in this study. The effects of clear aligners therapy on oral health related quality of life (OHRQoL) in comparison with vestibular fixed appliances using the validated OHIP-14 tool during orthodontic treatment. So the aim of the study was to compare the changes in OHRQoL between patients receiving clear aligners or fixed appliances during the first year of the orthodontic treatment.

There are two groups:

First group (Experimental): the patients in this group will be treated using clear aligners.

Second group (Control): the patients in this group will be treated using fixed appliances.

DETAILED DESCRIPTION:
For years, orthodontists and dentists have used removable appliances for orthodontic treatment. Today, with the CAD/CAM technology, clear aligners treat a broader range of cases with greater precision. They consists of a series of plastic aligners that are intended to replace conventional wire and bracket technology for many orthodontic cases. Each custom manufactured aligner exerts gentle, continuous forces to move teeth incrementally from their original state to a final, treated state. Each aligner is worn for about two weeks, then replaced by the next in the series until the final position is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Class I malocclusion with severe crowding (more than 5 mm of tooth-size-arch-length-discrepancy).
* Good oral hygiene and periodontal health.
* No congenitally missing or extracted teeth (except for the third molars).
* No history of previous trauma to the maxillofacial region or surgical interventions.

Exclusion Criteria:

* Previous orthodontic treatment.
* Subject with psychological abnormalities.
* Subject with systemic diseases.
* Subject has known allergy to latex and plastic

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Changes in oral health related quality of life | T0: immediately before the start of orthodontic treatment, T1: after 1 week, T2: after 2 weeks, T3: after 1 month, T4: after 6 months, T5: after 12 months
  Patients in both groups will be given a questionnaire to be filled. The questionnaire to be used is called Oral-Health-Impact-Profile with 14 items (OHIP-14) which can be filled in 3 minutes. OHIP-14 includes a subjective evaluation of the individual's oral health, functional well-being, emotional well-being, expectations and satisfaction with care and sense of self.

CONTACTS AND LOCATIONS:
Overall Officials: Samer T Jaber, DDS,MSc, Principal Investigator — PhD student at the Orthodontic Department, University of Damascus; Mohammad Y Hajeer, DDS,MSc,PhD, Study Chair — Associate Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azaripour A, Weusmann J, Mahmoodi B, Peppas D, Gerhold-Ay A, Van Noorden CJ, Willershausen B. Braces versus Invisalign(R): gingival parameters and patients' satisfaction during treatment: a cross-sectional study. BMC Oral Health. 2015 Jun 24;15:69. doi: 10.1186/s12903-015-0060-4. PMID 26104387
- [Background] Demirovic K, Habibovic J, Dzemidzic V, Tiro A, Nakas E. Comparison of Oral Health-Related Quality of Life in Treated and Non-Treated Orthodontic Patients. Med Arch. 2019 Apr;73(2):113-117. doi: 10.5455/medarh.2019.73.113-117. PMID 31391699
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Zhang B, Huang X, Huo S, Zhang C, Zhao S, Cen X, Zhao Z. Effect of clear aligners on oral health-related quality of life: A systematic review. Orthod Craniofac Res. 2020 Nov;23(4):363-370. doi: 10.1111/ocr.12382. Epub 2020 May 13. PMID 32340082
- [Background] Zhang M, McGrath C, Hagg U. The impact of malocclusion and its treatment on quality of life: a literature review. Int J Paediatr Dent. 2006 Nov;16(6):381-7. doi: 10.1111/j.1365-263X.2006.00768.x. PMID 17014535
- [Background] Zheng DH, Wang XX, Su YR, Zhao SY, Xu C, Kong C, Zhang J. Assessing changes in quality of life using the Oral Health Impact Profile (OHIP) in patients with different classifications of malocclusion during comprehensive orthodontic treatment. BMC Oral Health. 2015 Nov 20;15:148. doi: 10.1186/s12903-015-0130-7. PMID 26589825